CLINICAL TRIAL: NCT04946071
Title: Reducing HIV-Related Stigma in School Children in Northern Uganda: A Multi-level Arts-Based Population Health Intervention
Brief Title: Reducing HIV-related Stigma in School Children in Northern Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thompson Rivers University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The AIDS Support Organization (Other); Waroco Kwo Elders Association (Unknown); Omoro District Health Office (Unknown); Omoro District Education Office (Unknown)
Responsible Party: Principal Investigator, Bonnie Fournier, Associate Professor, Thompson Rivers University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 102240
Record Dates: First submitted 2021-05-28; First posted 2021-06-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: HIV-related Stigma; Health Risk Behaviors; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Health Risk Behaviors; Behavior

STUDY DESIGN:
Intervention Model Description: The study will employ a stepped-wedge, cluster randomized design involving crossover of clusters from the control to the intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Period in which each group will not receive the arts-based HIV stigma intervention.
- Group 1 (Experimental): Arts-based HIV stigma intervention for three 8-week periods (24 weeks). The intervention will begin with 5 weeks of two 2 interrelated activities: 1) Transformative educational activities that will engage learners in problem-based discussions; 2) Arts-based activities that will focus on addressing the "problem" through finding "solutions" and encouraging action will be accomplished by learning traditional Ugandan songs, dance, told and acted stories, proverbs and sayings that incorporate empowering messages and moral teachings connected with self and community, respect for self, peers and authority, and responsibility for others. These activities will be followed by 3 weeks of a participatory theatre intervention (PTI) developed by students that will summarize the learnings and cultural traditions from the weekly sessions.
  Interventions: Behavioral: Arts-based HIV stigma intervention
- Group 2 (Experimental): Arts-based HIV stigma intervention for two 8-week periods (16 weeks). Each intervention period will begin with 5 weeks of two 2 interrelated activities: 1) Transformative educational activities that will engage learners in problem-based discussions; 2) Arts-based activities that will focus on addressing the "problem" through finding "solutions" and encouraging action will be accomplished by learning traditional Ugandan songs, dance, told and acted stories, proverbs and sayings that incorporate empowering messages and moral teachings connected with self and community, respect for self, peers and authority, and responsibility for others. These activities will be followed by 3 weeks of a participatory theatre intervention (PTI) developed by students that will summarize the learnings and cultural traditions from the weekly sessions.
  Interventions: Behavioral: Arts-based HIV stigma intervention
- Group 3 (Experimental): Arts-based HIV stigma intervention for one 8-week period. The intervention period will begin with 5 weeks of two 2 interrelated activities: 1) Transformative educational activities that will engage learners in problem-based discussions; 2) Arts-based activities that will focus on addressing the "problem" through finding "solutions" and encouraging action will be accomplished by learning traditional Ugandan songs, dance, told and acted stories, proverbs and sayings that incorporate empowering messages and moral teachings connected with self and community, respect for self, peers and authority, and responsibility for others. These activities will be followed by 3 weeks of a participatory theatre intervention (PTI) developed by students that will summarize the learnings and cultural traditions from the weekly sessions.
  Interventions: Behavioral: Arts-based HIV stigma intervention

INTERVENTIONS:
Behavioral: Arts-based HIV stigma intervention — The intervention will consist of 2-hour weekly sessions offered to students in participating schools. HIV-related stigma will be addressed by providing key information related to HIV and stigma, facilitating the acquisition of coping skills, and utilizing local cultural practices facilitated by Elders using creative methods to shift existing social and cultural norms that produce and perpetuate stigmatization. Specific intervention activities will include three interrelated activities. The core 2-hour weekly session will cover (1) transformative educational activities; (2) arts-based activities; (3) a summative activity consisting of (3) participatory theatre activites.
  Arms: Group 1; Group 2; Group 3

SUMMARY:
Over 2.6 million children aged 0-15 years are living with HIV globally, with the majority living in low and middle income countries in sub-Saharan Africa. Addressing stigma associated with HIV is key given the significant harm that may be experienced in the form of negative health and social outcomes, reduced access to HIV prevention services, and increased vulnerability to infection. This stepped-wedge, cluster randomized trial with assess the impact of an arts-based HIV stigma intervention on knowledge and attitudes towards children who are HIV+ and - affected; enacted, internalized, anticipated, courtesy, and perceived stigma (primary outcomes); HIV testing frequency among sexually active participants; linkage to care, antiretroviral therapy (ART) initiation and adherence among HIV+ participants; and viral suppression among HIV+ participants (secondary outcomes) of children aged 10+ years in Omoro District, Uganda, post-intervention and 5-months post-intervention.

DETAILED DESCRIPTION:
Background: Over 2.6 million children aged 0-15 years are living with HIV globally, with the majority living in low and middle income countries in sub-Saharan Africa. Addressing stigma associated with HIV is key given the significant harm that may be experienced in the form of negative health and social outcomes, reduced access to HIV prevention services, and increased vulnerability to infection. Previous research among young people in Uganda showed that stigma is meted out in the form of verbal and physical abuse from teachers and peers (bullying), leading to social isolation, school drop-out, depression and suicidal ideation. Given the limited evidence available in support of effective stigma reduction among young people, efforts to help those affected constitute a major gap in the HIV prevention literature.

Purpose: The overall aim of the proposed study is to implement and evaluate an arts-based intervention rooted in local cultural knowledge to reduce stigma and improve HIV prevention outcomes among HIV positive and HIV- affected young people.

Methods: The study will employ a stepped-wedge, cluster randomized design involving crossover of clusters from the control to the intervention arm. The stepped-wedge design will consist of three groups (Group 1, Group 2, Group 3), each comprised of two primary and two secondary schools. Each time period will be 8 weeks in duration. Group 1 will receive the intervention for three time periods (24 weeks). Group 2 will receive the intervention over two time periods (16 weeks). Group 3 will receive the intervention over one time period (8 weeks). Formative qualitative interviews will also inform the arts-based HIV-stigma intervention and obtain additional data for research objectives. We will conduct at 50 qualitative semi-structured interviews, lasting between 30 minutes to 45 minutes, with purposively selected students, Elders, and teachers at participating schools. A community advisory committee (CAC) will inform all design elements and supervise implementation. Team members will collaborate to develop, implement, evaluate and disseminate results of the proposed study. Primary endpoints will include: 1) HIV stigma reduction; and, 2) knowledge increase. Secondary endpoints will include: 1) HIV testing frequency among sexually active participants; 2) linkage to care among HIV+ participants; 3) ART initiation among HIV+ participants; 4) ART adherence among HIV+ participants; and 5) viral suppression among HIV+ participants. Secondary endpoints will be measured through a local AIDS non-governmental organization (TASO) and the community health clinics who have agreed to provide access to their medical files. No blood samples will be drawn. Ages 10+ will participate in the study with parental consent.

Survey Data Analysis: Descriptive analyses will be used to describe clusters relative to their size at each time point (planned sample size and achieved sample size), key demographics and outcomes, and comparison of randomization groups. Main analyses will follow an intention-to-treat approach, with clusters analyzed as per original treatment assignment. Main analyses will use Linear Mixed Effect Models (LMEM) or Generalized Linear Mixed Effect Models (GLMEM) to assess the intervention effect. LMEM will be used for continuous outcomes that approach normality and GLMEM for binary and other types of outcomes. Normality will be assessed by the model residuals and outliers by Cook's Distance, Leverage and Residuals. Calendar time and school semester will be entered as fixed effects. The multilevel structure will be defined by participants as level 1 and clusters as level 2. All clustering levels will be specified as random effects. Sensitivity analyses will be performed of drop-outs and completers to better understand possible biases arising from attrition. A significance level of 0.05 will be used in all statistical tests.

Interview Data Analysis: Interviews will be coded using a constant-comparative and concept-development approach based on emergent themes that evolve throughout the course of the research. Initial coding will be done jointly by two researchers, and consensus negotiated. Matrix methodology techniques described by Miles, Huberman and Saldana will also be used in the analysis. First level analysis will be used to assign a descriptive code (label) to a segment of the data to give it meaning. As the researchers become more familiar with the data, pattern coding will be used to label emerging themes. An inductive approach will be used to analyze the data by iteratively coding and identifying themes and relationships between themes. Memos will be used to record methodological decisions and analytic insights. Validity will be assessed by convening focus groups for member checking the interpretation of data.

Significance: The study it will fill this evidence gap in HIV stigma intervention research and practice by creating and evaluating a transformative education and arts-based intervention using a participatory approach. The method of transforming cultural knowledge to an arts-based intervention may be a reproducible method for locally acceptable intervention design to improve HIV outcomes among young people.

ELIGIBILITY:
Inclusion Criteria:

* Children (age ≥10 years) in Omoro District, Northern Uganda
* Attending a government-funded primary and/or secondary school in the Omoro District
* Enrolled in primary grades 4-6 and secondary grades 1-3

Exclusion Criteria:

* Does not meet one or more inclusion criteria
* Those attending the following government-funded schools due to distance: Awere secondary school, Awere primary school, Dino primary school, Odek primary school, Agweno primary school, Jing Komi primary school, Acet primary school, Awali primary school, Aromo Wanglobo primary school, Binya primary school

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2900 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline and between time points in enacted, anticipated and internalized stigma towards HIV+ students | post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  measured using the Adolescents Living with HIV - Stigma Scale. The scale comprises of 10 items and will be administered by a member of the research team.
Change from baseline and between time points in courtesy stigma towards HIV+ students | post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  measured using the Brief Stigma by Association Scale in HIV-affected students. The scale comprises of 10 items and will be administered by a member of the research team.
Change from baseline and between time points in perceived stigma | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  measured using the Stewart's 10-item subscale on felt-normative stigma towards people living with HIV. The scale will be administered by a member of the research team.
Change from baseline and between time points in HIV knowledge | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  measured using questionnaire on HIV knowledge. Questionnaire will be administered by a member of the research team.
Change from baseline and between time points for fear of HIV transmission and disease | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  measured using questionnaire on fear of HIV transmission and disease. Questionnaire will be administered by a member of the research team.

SECONDARY OUTCOMES:
HIV testing frequency among sexually active participants | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  HIV confirmation/diagnosis dates and HIV status. Review of personal health records from community health clinics, and individual medical variables will be crossed-referenced with survey responses, with authorization from the participant (children 13-18 years) and guardian/parent (children 10-12 years).
Initiation of linkage to care among HIV+ participants | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  Initiation of linkage to care (yes/no) through review of personal health records from community health clinics and individual medical variables will be crossed-referenced with survey responses, with authorization from the participant and guardian/parent.
ART initiation among HIV+ participants | Baseline (0 weeks), post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  Initiation of ART initiation (yes/no) through review of personal health records from community health clinics and individual medical variables will be crossed-referenced with survey responses, with authorization from the participant and guardian/parent.
Change from baseline and between time points in viral suppression among HIV+ participants | post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  copies/ml, through review of personal health records from community health clinics with authorization from the participant and guardian/parent.
Change from baseline and between time points in ART adherence | post-intervention (8 weeks), post-intervention (16 weeks), post-intervention (24 weeks), 5 months post-intervention.
  capsules taken/capsules prescribed, through review of personal health records from community health clinics and individual medical variables will be crossed-referenced with survey responses, with authorization from the participant and guardian/parent.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Fournier, PhD RN, Principal Investigator — Thompson Rivers University
Locations (1):
- Omoro District, Palenga, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendelsohn JB, Fournier B, Caron-Roy S, Maina G, Strudwick G, Ojok S, Lim HJ, Sanches M, Logie CH, Sommerfeldt S, Nykiforuk C, Harrowing J, Adyanga FA, Hakiigaba JO, Bilash O. Reducing HIV-related stigma among young people attending school in Northern Uganda: study protocol for a participatory arts-based population health intervention and stepped-wedge cluster-randomized trial. Trials. 2022 Dec 23;23(1):1043. doi: 10.1186/s13063-022-06643-9. PMID 36564802